CLINICAL TRIAL: NCT07351084
Title: Retrospective Chart Review Study of Patient Factors Associated With Fragmentation of Copper Intrauterine Devices Requiring Hysteroscopic Removal
Brief Title: Patient Factors Associated With Fragmentation of Copper Intrauterine Devices Requiring Hysteroscopic Removal
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00160745
Record Dates: First submitted 2026-01-09; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-08

CONDITIONS: Intrauterine Device Complications; Contraceptive Device Failure; IUD Fragmentation; Retained Intrauterine Device; Female Contraception; Women's Health; Reproductive Health
Keywords: Copper IUD; ParaGard; Intrauterine device; IUD breakage; IUD retention; IUD complications; Hysteroscopy; IUD removal; IUD fracture; Gynecologic surgery; Contraception complications; Retained IUD fragment; Minimally invasive gynecology; Long-acting reversible contraception (LARC)
MeSH Terms: interventions — Hysteroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hysteroscopy: Necessitated a hysteroscopic procedure.
  Interventions: Other: Hysteroscopy

INTERVENTIONS:
Other: Hysteroscopy — Retrospective chart review for those patients who had a hysteroscopy after IUD removal.

SUMMARY:
The purpose of this retrospective chart review was to identify risks factors for patients associated to Cooper IUD fragmentation upon removal resulting in the requirement of a hysteroscopy evaluation.

ELIGIBILITY:
Inclusion Criteria:

* IUD removal and required hysteroscopy

Exclusion Criteria:

* Younger than 18 years old
* IU removal without requiring hysteroscopy

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Study Population: Patients who underwent IUD removal at the University of Kansas Health System
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Hysteroscopy Resulting from IUD Fragmentation Upon Removal | 2005-2025
  Identify patient risk factors for Cooper IDU fragmentation upon removal requiring a hysteriscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Annabel Mancillas, MD MPH FACOG, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States